CLINICAL TRIAL: NCT03686098
Title: The Malaysian Soy and Mammographic Density (MiSo) Study: A Randomized, Three-arm, Controlled Clinical Trial to Investigate the Impact of Soy Isoflavone Intake on Mammographic Density as a Biomarker of Breast Cancer Risk
Brief Title: The Malaysian Soy and Mammographic Density Study
Acronym: MiSo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cancer Research Malaysia (Other)
Collaborators: University of Nottingham Malaysia (Other); Subang Jaya Medical Centre (Unknown); Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRM-BRE-002
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer; Mammographic Density
Keywords: Diet; Soy; Prevention; Asian; Breast Cancer; Mammographic Density; Isoflavones
MeSH Terms: conditions — Breast Neoplasms | interventions — Soybean Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dietary Soy Arm (Experimental): Participants will be asked to increase soy in their diet by an equivalent of 50mg/day for 12 months
  Interventions: Dietary Supplement: Dietary soy
- Soy Supplement Arm (Active Comparator): Participants will consume 2 tablets of 50mg each per day for 12 months
  Interventions: Dietary Supplement: Soy Supplement
- Control Arm (No Intervention): No diet or supplement changes

INTERVENTIONS:
Dietary Supplement: Dietary soy — Soy isoflavones delivered through diet, assisted by a detailed food guide for locally available soy-based foods.
  Arms: Dietary Soy Arm
Dietary Supplement: Soy Supplement — Soy isoflavones delivered in extracted form
  Arms: Soy Supplement Arm

SUMMARY:
Globally, breast cancer is the most common cancer and the main cause of deaths due to cancer. This is attributed to changes in reproductive habits as well as an increasingly sedentary lifestyle, with low physical activity and diets rich in saturated fats but low in fiber. While the main focus in many Asian countries is to improve survival from breast cancer by encouraging early detection of the disease and improving access to cancer treatment, it does not reduce the number of women who will be diagnosed with breast cancer in the years to come. Currently, there is an urgent need to develop effective strategies to prevent breast cancer in Asia and beyond.

Soy may be an important dietary strategy for breast cancer prevention. Compared to women in the West, Asian women consume up to 10-fold more soy in their diet, which may, in part, explain their lower risk of breast cancer. Soybeans are rich in isoflavones, which can mimic estrogenic activity. In the body, it competes with estrogen and binds to estrogen receptor sites, thereby reducing the effect of estrogen and possibly lowering breast cancer risk.

Consistently, research has shown that Asian postmenopausal women who have high soy diets are less likely to be diagnosed with breast cancer. However, researchers have not been able to show that postmenopausal women can reduce their breast cancer risk by increasing soy intake as part of their diets. There are several reasons why these studies have failed to see an effect despite the body of evidence indicating that soy may be protective. Firstly, these are studies of Caucasian women who may have never been exposed to soy, particularly in adolescence, where soy may have the greatest impact. Also, these studies have used soy isoflavone supplements, rather than traditional soy foods made from whole soybeans, which may affect how soy is metabolized in the body. Lastly, the way in which mammographic density measurements were obtained previously could have negatively influenced the study results, such as the use of digitized images of mammogram films rather than raw digital images and the use of semi-automated methods that may be subject to human error and reader variability.

Therefore, a well-designed intervention study among Asian women living in Asia, using suitable mammographic density measures as a surrogate marker of breast cancer risk, will best answer these remaining gaps in our knowledge about the soy-breast cancer relationship.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Malaysian Mammography Study and agreed to be contacted
* Aged between 45 and 65 years old at study recruitment (i.e. as of June 2018)
* No genetic predisposition to breast cancer (carriers of the BRCA1 and BRCA2 mutations)
* Measurable amount of mammographic density (at least 4.5% Volpara percent mammographic density).

Exclusion Criteria:

* Personal history of breast cancer
* Personal history of other cancers, stroke, and other serious health conditions
* Personal history of benign breast disease
* Pre-menopausal (regular menstrual periods) or early peri-menopausal women (irregular menstrual period with a menstrual period in the past 3 months)
* Women who have a history of high uric acid, gout and associated conditions
* Women who have been diagnosed as diabetic or pre-diabetic
* Women who have been diagnosed with hypothyroidism
* Women who have gastrointestinal conditions (i.e. irritable bowel syndrome)
* Women who are allergic or intolerant to soy and soy products
* Currently (within the last 6 months) on hormone replacement therapy drugs, including alternative and traditional therapies for menopause symptom management
* Currently (within the last 6 months) a smoker
* Women who report a high soy diet (consuming soy foods at least once a day or are currently taking soy supplements
* Women who have had a mammogram in the past 12 months
* Women with breast augmentation
* Women with an abnormal or suspicious mammogram at recruitment. This includes women who are scored 2-5 using American College of Radiology's BIRADS (Version 5), unless reported as normal after additional tests (i.e. ultrasound). For women with dense breast, we will exclude women with an abnormal ultrasound (indicative of benign or malignant disease).

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2018-11-19 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Mammographic Density | 12 months
  Measurement of change in mammographic density over the study period

CONTACTS AND LOCATIONS:
Overall Officials: Soo Hwang Teo, Principal Investigator — Cancer Research Malaysia
Locations (1):
- Cancer Research Malaysia, Subang Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rajaram N, Yap B, Eriksson M, Mariapun S, Tan LM, Sa'at H, Ho ELM, Taib NAM, Khor GL, Yip CH, Ho WK, Hall P, Teo SH. A Randomized Controlled Trial of Soy Isoflavone Intake on Mammographic Density among Malaysian Women. Nutrients. 2023 Jan 6;15(2):299. doi: 10.3390/nu15020299. PMID 36678170
- See also: Official website of Cancer Research Malaysia — http://www.cancerresearch.my